CLINICAL TRIAL: NCT03118466
Title: Phase 2 Study of Mitoxantrone, Etoposide, and Cytarabine (MEC) Plus Lenalidomide for the Treatment of Adult Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Mitoxantrone, Etoposide, and Cytarabine (MEC) Plus Lenalidomide for Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Andrew Mark Brunner, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-574
Record Dates: First submitted 2017-03-30; First posted 2017-04-18 (Actual); Results first posted 2021-02-03 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: AML
Keywords: AML
MeSH Terms: interventions — Etoposide; Cytarabine; Lenalidomide; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide and MEC chemotherapy (Experimental): Lenalidomide is taken orally on a daily basis days 1-10. Mitoxantrone, Etoposide, and Cytarabine are administered intravenously on a daily basis for days 4 through 8 of the treatment. There is only one cycle of treatment in this study.
  Interventions: Drug: Etoposide; Drug: Cytarabine; Drug: Lenalidomide; Drug: Mitoxantrone

INTERVENTIONS:
Drug: Etoposide — A Drug that interfere with the action of topoisomerase enzymes (topoisomerase I and II). Topoisomerase enzymes control the manipulation of the structure of DNA necessary for replication.
  Other Names: Toposar
Drug: Cytarabine — Cytarabine is an antimetabolite antineoplastic agent that inhibits the synthesis of DNA.
  Other Names: Depocyt
Drug: Lenalidomide — It may act by inhibiting the growth of new blood vessels (angiogenesis) in tumors, enhancing the status of the immune system, or decreasing cytokine and growth factor production
  Other Names: REVLIMID
Drug: Mitoxantrone — It interfere with cell reproduction
  Other Names: Novantrone

SUMMARY:
This research study is evaluating how a drug called lenalidomide, given in combination with the standard chemotherapy regimen of Mitoxantrone, Etoposide, and Cytarabine, commonly referred to as MEC, works in individuals with either relapsed or refractory AML

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved lenalidomide for this specific disease, but it has been approved for other uses, including for patients with multiple myeloma and some patients with myelodysplastic syndrome. This treatment is investigational because it is not approved by the FDA for patients with AML. Lenalidomide is a chemotherapy that also modulates the immune system, and is in a category of drugs called immunomodulatory drugs or IMIDs. Some research studies suggest that lenalidomide may be effective in patients with AML. Since the investigators know that many patients who receive MEC chemotherapy alone have less than desired response rates and overall shorter periods of remission (time free from leukemia) after treatment, the investigators are studying whether the addition of lenalidomide to MEC improves upon typical responses.

The combination of MEC (mitoxantrone, etoposide, and cytarabine) is a standard treatment option, commonly used for relapsed or refractory acute myeloid leukemia.

.

ELIGIBILITY:
Inclusion Criteria:

* Acute myelogenous leukemia diagnosed by WHO criteria with one of the following (patients with biphenotypic leukemia are eligible, provided that the treating physician determines an AML treatment regimen is appropriate)

  * Primary refractory disease following > 1cycle of chemotherapy, (such as hypomethylating agent or induction chemotherapy)
  * First relapse or higher. Patients with primary or secondary acute myelogenous leukemia are eligible.
* Age 18-70 years old
* LVEF > 50 %
* ECOG Performance status 0-2
* Able to adhere to study schedule and other protocol requirements.
* Participants must have normal organ function as defined below, unless felt due to underlying disease and approved by the overall PI. Patients with Gilbert's disease may have total bilirubin up to < 3 x ULN.

  * Creatinine < 2.0mg/dl
  * Total bilirubin < 1.5 x ULN
  * AST (SGOT) and ALT (SGPT) < 3 x ULN.
* Patients may receive hydroxyurea, steroids, or leukapheresis as necessary until Day 5 of treatment.
* Patients must give voluntary written informed consent and HIPAA authorization before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Patients may have had prior treatment for MDS or AML, including prior lenalidomide for MDS or AML or another condition.
* Patient may have had prior autologous or allogeneic transplant (family member, unrelated donor, or cord blood) if there is at least 90 days between transplant and study entry.
* Patients may also have had donor lymphocyte infusion if there is at least 60 days between donor lymphocyte infusion and study entry.
* Patients on immunosuppression are also eligible.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL prior to receiving treatment with lenalidomide, and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
* Ability to understand and the willingness to sign a written informed consent document.
* All study participants must be registered into the mandatory Revlimid REMS ® program, and be willing and able to comply with the requirements of the REMs ® program. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program

Exclusion Criteria:

* Known hypersensitivity to thalidomide or lenalidomide (if applicable).
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Known seropositive for human immunodeficiency virus (HIV). HIV testing is not required. Hepatitis testing is not required.
* Patients who have had a myocardial infarction within 6 months of enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Any serious medical condition laboratory abnormality or psychiatric illness that would prevent the subject from signing the consent form.
* Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Patients with major surgery within 28 days prior to treatment.
* Patients with any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Patient has received an investigational agent or cytotoxic chemotherapy (excluding hydroxyurea) within 7 days of study entry.
* Patients with acute promyelocytic leukemia.
* Females who are pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2021-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Brunner, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts general Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient came off study prior to receiving any treatment and was replaced. A total of 40 patients received study treatment.
Period: Overall Study
Arm/Group | Lenalidomide and MEC chemotherapy
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide and MEC chemotherapy
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 56 [19 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Percentage of patients who have achieve CR or CRp after treatment.
  * Morphologic Complete Remission (CR): Defined as morphologic leukemia-free state, including <5% blasts in Bone Marrow aspirate with marrow spicules, no persistent extramedullary disease, ANC >1000/mm3 and platelet count >100,000/mm3.
  * Morphologic Complete Remission without platelet recovery (CRp): Defined as CR with the exception of platelet count < 100,000/mm3 (CRp).
Time Frame: up to 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide and MEC chemotherapy
Number analyzed (Participants) | 40
Participants | 19

2. Secondary Outcome: Number of Patients That Achieved ANC Recovery
Description: The number of patients that achieved a neutrophil count of > 500/mm3 for 3 days within 45 of starting treatment
Time Frame: up to 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide and MEC chemotherapy
Number analyzed (Participants) | 40
Participants | 25

3. Secondary Outcome: Number of Patients That Achieved Platelet Recovery
Description: The number of patients that achieved a stable platelet count > 20,000/mm3 for 3 days within 45 days of starting treatment
Time Frame: up to 45 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide and MEC chemotherapy
Number analyzed (Participants) | 40
Participants | 27

4. Secondary Outcome: Treatment-related Mortality
Description: Cumulative number of deaths not related to persistent or relapsed leukemia during treatment within 50 days of the start of treatment.
Time Frame: 50 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide and MEC chemotherapy
Number analyzed (Participants) | 40
Participants | 2

5. Secondary Outcome: Transfusion Support: Number of Red Blood Cell and Platelet Transfusions
Description: Number of red blood cell and platelet transfusions received within the first 50 days of treatment
Time Frame: 50 days
Measure: Median (Full Range); unit: Number of Transfusions
Arm/Group | Lenalidomide and MEC chemotherapy
Number analyzed (Participants) | 40
Number of Transfusions
  Platelet Transfusions | 7 [2 to 49]
  Red Blood Cell Transfusions | 9 [1 to 47]

6. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from diagnosis of disease until date of death or censored on the last known date alive if patients are still alive.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide and MEC chemotherapy
Number analyzed (Participants) | 40
Months | 16 [13 to NA] — Upper limit of confidence interval not defined due to insufficient number of events

7. Secondary Outcome: Relapse-Free Survival
Description: Relapse-Free Survival is defined as time from diagnosis of disease until date of relapse, death, or censored on the last known date alive if patients are still alive.Relapse is defined by morphological evidence of the original malignancy consistent with pre-treatment features.
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide and MEC chemotherapy
Number analyzed (Participants) | 40
months | 13.1 [10.2 to NA] — 95% CI is 10.2 - NR; Upper limit of confidence interval not defined due to insufficient number of events

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the end of study treatment, up to 3 years
Arm/Group | Lenalidomide and MEC chemotherapy
All-Cause Mortality (participants affected / at risk) | 15/40
Serious Adverse Events (participants affected / at risk) | 19/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and MEC chemotherapy (N=40)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (5)
Abdominal infection (Infections and infestations) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (3)
Infections and infestations - Other, candidemia sepsis (Infections and infestations) | 1 (1)
Infections and infestations - Other, Enterococcus faecium bacteremia (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and MEC chemotherapy (N=40)
Anemia (Blood and lymphatic system disorders) | 20 (33)
Febrile neutropenia (Blood and lymphatic system disorders) | 27 (37)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 5 (7)
Chills (General Disorders) | 5 (5)
Edema face (General Disorders) | 4 (5)
Edema limbs (General Disorders) | 15 (17)
Fatigue (General Disorders) | 20 (25)
Fever (General Disorders) | 16 (21)
Malaise (General Disorders) | 3 (3)
Non-cardiac chest pain (General Disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (22)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 11 (21)
Bloating (Gastrointestinal disorders) | 2 (3)
Colitis (Gastrointestinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 10 (12)
Diarrhea (Gastrointestinal disorders) | 22 (31)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 2 (2)
Esophageal pain (Gastrointestinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Gingival pain (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 7 (9)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 10 (12)
Nausea (Gastrointestinal disorders) | 22 (27)
Oral pain (Gastrointestinal disorders) | 4 (5)
Rectal pain (Gastrointestinal disorders) | 5 (10)
Typhlitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 12 (14)
Catheter related infection (Infections and infestations) | 5 (5)
Lung infection (Infections and infestations) | 6 (7)
Skin infection (Infections and infestations) | 4 (4)
Alanine aminotransferase increased (Investigations) | 11 (21)
Alkaline phosphatase increased (Investigations) | 5 (9)
Aspartate aminotransferase increased (Investigations) | 10 (16)
Blood bilirubin increased (Investigations) | 8 (17)
Creatinine increased (Investigations) | 3 (3)
INR increased (Investigations) | 3 (5)
Lymphocyte count decreased (Investigations) | 3 (6)
Neutrophil count decreased (Investigations) | 12 (21)
Platelet count decreased (Investigations) | 22 (63)
Weight loss (Investigations) | 3 (8)
White blood cell decreased (Investigations) | 5 (10)
Anorexia (Metabolism and nutrition disorders) | 18 (29)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (10)
Hypokalemia (Metabolism and nutrition disorders) | 13 (38)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (7)
Hyponatremia (Metabolism and nutrition disorders) | 6 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 14 (30)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal and connective tissue disorder - (Musculoskeletal and connective tissue disorders) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 9 (11)
Dysgeusia (Nervous system disorders) | 4 (5)
Headache (Nervous system disorders) | 10 (13)
Paresthesia (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 4 (4)
Blurred vision (Eye disorders) | 4 (4)
Dry eye (Eye disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 6 (6)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 11 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hematuria (Renal and urinary disorders) | 3 (3)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (3)
Flushing (Vascular disorders) | 3 (3)
Hematoma (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 17 (22)
Thromboembolic event (Vascular disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT03118466/Prot_SAP_000.pdf